CLINICAL TRIAL: NCT02236754
Title: Scan Re-Scan Pancreatic Beta Cell Imaging Using PET Imaging and 18 F-FP-DTBZ
Brief Title: Evaluation of 18 F-FP-DTBZ Pancreatic PET Scanning as a Tool to Measure Beta Cell Mass
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAAJ5709; R01DK077493-03 (NIH)
Record Dates: First submitted 2014-01-28; First posted 2014-09-11 (Estimated); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers; Diabetes Mellitus, Type 1
Keywords: dihydrotetrabenazine; beta cell mass; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — florbenazine F 18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Controls (Other): Pancreatic 18 F-FP-DTBZ uptake will be measured with PET scanning in healthy controls: subjects with predicted normal BCM (healthy, normal weight, non-diabetic individuals who have stimulated insulin and c-peptide levels within the normal range).
  Interventions: Drug: 18 F-FP-DTBZ; Radiation: PET Scanning
- Patients with T1D (Other): Pancreatic 18 F-FP-DTBZ uptake will be measured with PET scanning in patients with longstanding T1D: subjects with predicted reduced beta cell mass (subjects with established T1DM who have low or no measurable stimulated insulin and c-peptide levels).
  Interventions: Drug: 18 F-FP-DTBZ; Radiation: PET Scanning

INTERVENTIONS:
Drug: 18 F-FP-DTBZ — The drug, no carrier added [18 F]-FP-DTBZ, is formulated in 5% (v/v) ethanol in 0.9% sterile saline solution to produce [18 F]-FP-DTBZ for injection. Subjects will receive a single i.v. administration of no more than 7.6 millicuries (mCi) of [18 F]-FP-DTBZ for injection immediately prior to imaging. The specific activity at time of injection will less than 1.0 mCi/microgram and thus for a 7.6 mCi dose the maximal mass dose will be less than 10 microgram.
Radiation: PET Scanning — Individuals will be imaged continuously (i.e. dynamically) for 2 hours.
  Other Names: Positron Emission Tomography

SUMMARY:
Type 1 diabetes mellitus (T1DM) develops when there is impaired insulin production due to loss of insulin producing cells (beta cells). The amount of insulin that can be produced is imperfectly correlated with beta cell mass (BCM). The development of a reliable method to noninvasively quantify the total amount of insulin producing beta cells would be of great benefit by providing an important endpoint for the development of new treatments of diabetes. The investigators have previously identified a specific marker on islet cells called vesicular monoamine transporter 2 (VMAT2) that the investigators now propose to use in positron emission tomography (PET) scanning to determine islet beta cell mass. The PET radiopharmaceutical 18 F-fluoropropyl(FP)-dihydrotetrabenazine(DTBZ) has been used previously in human subjects without adverse effects. It has shown promise in differentiating type 1 diabetes and non-diabetes. The investigators now hypothesize that repeat PET scans will be reproducible in the same subject. Subjects with normal BCM will be recruited from among normal weight non-diabetic people with plasma insulin levels within the normal range. Subjects with predicted reduced BCM will be recruited from among patients with T1DM who have low or non-measurable insulin levels. Two PET scan measurements will be taken in each subject and the amount of VMAT2 in the pancreas will be and compared for reproducible findings. Biochemical testing will also be performed and compared to PET scans as a potential indirect marker of beta cell mass.

DETAILED DESCRIPTION:
Diabetes results when the insulin secretory capacity of the beta cell population is lost or severely compromised.Plasma insulin levels have been used as a surrogate marker of beta cell mass (BCM) but insulin levels often do not correlate well. A "gold standard of measurement" to obtain BCM would be of great value. The aim of the proposed study is to evaluate an islet imaging technique using PET scanning to directly measure BCM and thus provide valuable information for monitoring disease progress and response to therapy in people with diabetes and in people at high risk for diabetes. Type 1 diabetes (T1DM) occurs when the beta cells are selectively destroyed by a T cell mediated autoimmune process. People at high risk for developing T1DM, such as first degree relatives of patients with T1DM, can sometimes be identified before the disease develops by measuring autoantibodies to beta cells, however this test is neither sensitive nor specific. Little is known about the natural history of BCM, turnover and cell lifetime, or the course of inflammation in diabetes. This is principally because the pancreas is a highly heterogeneous organ that is difficult to biopsy without significant complications, and BCM only comprises 1 to 2% of the total volume. Accurate assessment of BCM in human diabetes is limited to autopsy studies, which usually suffer from inadequate clinical information; thus, the development of non-invasive means of BCM measurement could be important for interventional therapies of T1DM, islet regeneration/stem cell therapy and islet transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes may be enrolled if they meet all of the following criteria:

  1. Are males or females between 18 and 70 years of age, inclusive
  2. Have a diagnosis of type 1 diabetes mellitus as defined by the American Diabetes Association (ADA) criteria or by diagnosed as per their endocrinologist; duration >5 years; Insulin dose requirements <0.8 units/kg/day
  3. HbA1c level between 5% and 8.5%
  4. Have fasting C-Peptide < 0.1 ng/ml
  5. Have a body mass index (BMI) between 18 and 32 kg/m2
  6. Able to tolerate PET imaging
  7. In the judgment of the physician, are capable of fasting 4 to 6 hours prior to screening and Day 1 imaging procedures
  8. Give informed consent

Healthy volunteers may be enrolled if they meeting all of the following criteria:

1. Are males or females between 18 and 70 years of age, inclusive
2. Have no history of type 1 or type 2 diabetes in a first degree relative
3. Fasting blood glucose less than 100 mg/dL
4. HbA1c level less than 6%
5. Normal Mixed Meal Tolerance test at screening visit
6. BMI between 18 and 32 kg/m2
7. Able to tolerate PET imaging
8. In the judgment of the physician, are capable of fasting 4 to 6 hours prior to screening and Day 1 imaging procedures, and
9. Give informed consent

Exclusion Criteria:

* Potential participants must not have any of the following exclusion criteria:

  1. Clinically significant renal dysfunction
  2. Clinically significant liver dysfunction as determined by history, physical examination, and standard liver function testing at screening (aspartate aminotransferase (AST), alanine aminotransferase (ALT), Total/Direct Bilirubin, Alkaline Phosphatase)
  3. Coagulopathy
  4. Use medications known to affect dopaminergic function, including monoamine oxidase (MAO) inhibitors, tetrabenazine, or levodopa
  5. Recent (within 3 months) or current treatment with drugs influencing beta cell function or insulin sensitivity (e.g. glucocorticoids, reserpine) medications known to affect dopaminergic function, including MAO inhibitors, tetrabenazine, or levodopa
  6. Have polycystic ovarian syndrome
  7. History of movement disorder such as Parkinson's Disease, Huntington's Disease
  8. Clinically significant psychiatric disease or history of psychiatric illness such as depression, bipolar disease, anxiety or schizophrenia
  9. Current use (within past year) of cocaine, methamphetamine, and/or ecstasy (3,4methylenedioxymethamphetamine (MDMA))
  10. Have a recent history of alcohol or substance abuse or dependence
  11. Clinically significant cardiovascular disease or clinically significant abnormalities on screening electrocardiogram (ECG) (including but not limited to QT-interval time corrected > 450 msec)
  12. Clinically significant pulmonary, renal or hepatic impairment, or cancer
  13. Have clinically significant infectious disease, including acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV) infection or previous positive test for hepatitis B, hepatitis C, or HIV.
  14. Are women of childbearing potential not refraining from sexual activity or not using adequate contraception.

      Women must not be pregnant (negative serum human chorionic gonadotropin (hCG) at the time of screen) or breastfeeding at screening, and must agree to take appropriate steps not to become pregnant during for 30 days following the clinical trial
  15. Require medications with a narrow therapeutic window (e.g., warfarin), are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days
  16. Weigh more than the manufacturer recommended limit for the PET/computed tomography (CT) camera being used
  17. Any prior participation in other research protocols within the past month that involved radiation, with the exception of plain radiography studies (i.e., chest x-rays); And
  18. Have received a diagnostic or therapeutic radiopharmaceutical within the past week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2014-04-23 (Actual); Study Completion 2014-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harris, PhD, Principal Investigator — Columbia University
Locations (1):
- Naomi Berrie Diabetes Center, New York, New York, United States

REFERENCES:
- [Background] Goland R, Freeby M, Parsey R, Saisho Y, Kumar D, Simpson N, Hirsch J, Prince M, Maffei A, Mann JJ, Butler PC, Van Heertum R, Leibel RL, Ichise M, Harris PE. 11C-dihydrotetrabenazine PET of the pancreas in subjects with long-standing type 1 diabetes and in healthy controls. J Nucl Med. 2009 Mar;50(3):382-9. doi: 10.2967/jnumed.108.054866. Epub 2009 Feb 17. PMID 19223416
- [Result] Freeby MJ, Kringas P, Goland RS, Leibel RL, Maffei A, Divgi C, Ichise M, Harris PE. Cross-sectional and Test-Retest Characterization of PET with [(18)F]FP-(+)-DTBZ for beta Cell Mass Estimates in Diabetes. Mol Imaging Biol. 2016 Apr;18(2):292-301. doi: 10.1007/s11307-015-0888-7. Epub 2015 Sep 14. PMID 26370678
- See also: Investigator web site — http://www.nbdiabetes.org/news/using-nuclear-imaging-measure-beta-cell-mass-and-function

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects with diabetes were recruited at the Naomi Berri Diabetes Center. The physician ascertained from the patient that he/she is willing to discuss the study with the research team before the investigators approach the patient. Non-diabetic subjects were either be referred by their physicians, by word of mouth, or by flyer.
Groups:
- Healthy Controls: Pancreatic 18 F-FP-DTBZ uptake will be measured with positron emission tomography (PET) scanning in healthy controls: subjects with predicted normal beta cell mass (BCM) (healthy, normal weight, non-diabetic individuals who have stimulated insulin and c-peptide levels within the normal range).
  18 F-FP-DTBZ: The drug, no carrier added [18 F]-Fluoropropyl (FP)- dihydrotetrabenazine (DTBZ), is formulated in 5% (v/v) ethanol in 0.9% sterile saline solution to produce [18 F]-FP-DTBZ for injection. Subjects will receive a single i.v. administration of no more than 7.6 millicurie (mCi) of [18 F]-FP-DTBZ for injection immediately prior to imaging. The specific activity at time of injection will less than 1.0 mCi/microgram and thus for a 7.6 mCi dose the maximal mass dose will be less than 10 microgram.
  PET Scanning: Individuals will be imaged continuously (i.e. dynamically) for 2 hours.
- Patients With T1D: Pancreatic 18 F-FP-DTBZ uptake will be measured with PET scanning in patients with longstanding Type 1 Diabetes Mellitus (T1DM): subjects with predicted reduced beta cell mass (subjects with established T1DM who have low or no measurable stimulated insulin and c-peptide levels).
  18 F-FP-DTBZ: The drug, no carrier added [18 F]-FP-DTBZ, is formulated in 5% (v/v) ethanol in 0.9% sterile saline solution to produce [18 F]-FP-DTBZ for injection. Subjects will receive a single i.v. administration of no more than 7.6 mCi of [18 F]-FP-DTBZ for injection immediately prior to imaging. The specific activity at time of injection will less than 1.0 mCi/microgram and thus for a 7.6 mCi dose the maximal mass dose will be less than 10 microgram.
  PET Scanning: Individuals will be imaged continuously (i.e. dynamically) for 2 hours.
Period: Overall Study
Arm/Group | Healthy Controls | Patients With T1D
Started | 15 | 8
Completed | 14 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls: Pancreatic 18 F-FP-DTBZ uptake will be measured with PET scanning in healthy controls: subjects with predicted normal BCM (healthy, normal weight, non-diabetic individuals who have stimulated insulin and c-peptide levels within the normal range).
  18 F-FP-DTBZ: The drug, no carrier added [18 F]-FP-DTBZ, is formulated in 5% (v/v) ethanol in 0.9% sterile saline solution to produce [18 F]-FP-DTBZ for injection. Subjects will receive a single i.v. administration of no more than 7.6 mCi of [18 F]-FP-DTBZ for injection immediately prior to imaging. The specific activity at time of injection will less than 1.0 mCi/microgram and thus for a 7.6 mCi dose the maximal mass dose will be less than 10 microgram.
  PET Scanning: Individuals will be imaged continuously (i.e. dynamically) for 2 hours.
- Patients With T1D: Pancreatic 18 F-FP-DTBZ uptake will be measured with PET scanning in patients with longstanding T1D: subjects with predicted reduced beta cell mass (subjects with established T1DM who have low or no measurable stimulated insulin and c-peptide levels).
  18 F-FP-DTBZ: The drug, no carrier added [18 F]-FP-DTBZ, is formulated in 5% (v/v) ethanol in 0.9% sterile saline solution to produce [18 F]-FP-DTBZ for injection. Subjects will receive a single i.v. administration of no more than 7.6 mCi of [18 F]-FP-DTBZ for injection immediately prior to imaging. The specific activity at time of injection will less than 1.0 mCi/microgram and thus for a 7.6 mCi dose the maximal mass dose will be less than 10 microgram.
  PET Scanning: Individuals will be imaged continuously (i.e. dynamically) for 2 hours.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Patients With T1D | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 8 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean VMAT2 Functional Binding Capacity in the β Cells to 18 F-FP-DTBZ
Description: The VMAT2 functional binding capacity in the body and tail of the pancreas is calculated as BPND (VMAT2 binding potential) × PET ROI (region-of-interest) Volume. BPND is unitless, and ROI unit is mL. Higher values of the VMAT functional binding capacity indicates greater β cell mass.
Time Frame: Up to 2 months from enrollment
Measure: Mean (Standard Error); unit: unitless
Groups:
- Study Controls: Healthy individuals with no familial history of diabetes
- Longstanding T1D: Patients with Type 1 diabetes of duration longer than 5 years
Arm/Group | Study Controls | Longstanding T1D
Number analyzed (Participants) | 14 | 8
unitless | 103 (12) | 38 (5)

ADVERSE EVENTS:
Time Frame: Throughout study period, up to 2 months
Arm/Group | Study Controls | Longstanding T1D
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 0/14 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No